CLINICAL TRIAL: NCT03058458
Title: A First-time-in-human, Randomised, Double-blind, Placebo-controlled, Parallel-group Study in Healthy Volunteers and Patients With Asthma to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending and Repeat Doses of PIN201104
Brief Title: A First Time in Human Study of PIN201104 in Healthy Volunteers and Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peptinnovate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1104-001
Record Dates: First submitted 2017-01-24; First posted 2017-02-23 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD PIN201104 in Healthy Volunteers (HV) (Experimental): PIN201104 or placebo IV administration, single dose, 10 dose cohorts
  Interventions: Drug: PIN201104; Drug: Placebo
- Repeat dose PIN201104 in HV (Experimental): PIN201104 or placebo IV administration, 3 doses on single day, 1 cohort
  Interventions: Drug: PIN201104; Drug: Placebo
- Single dose PIN201104 in asthma patients (Experimental): PIN201104 or placebo IV administration, single dose, 2 cohorts
  Interventions: Drug: PIN201104; Drug: Placebo
- Single SC dose in HV (Experimental): PIN201104 or placebo SC administration, single dose, 1 cohort
  Interventions: Drug: PIN201104; Drug: Placebo

INTERVENTIONS:
Drug: PIN201104 — IV or SC administration
Drug: Placebo — IV or SC administration

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of different single and repeat doses of PIN201104 in healthy volunteers and in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects of non-childbearing potential age 18 to 65 years of age, and in good health as determined by medical history, physical examination, vital signs, electrocardiogram, and laboratory tests.
* Written informed consent must be obtained before any assessment is performed.
* Able to communicate well with the Investigator/designee.

Exclusion Criteria:

* Any known reaction to study drug or components
* concurrent or recent infection or clinically significant conditions that may place subject at risk or interference with absorption, distribution or excretion of drugs
* No QTcF interval ≥450 milliseconds, no QRS complex ≥120 milliseconds, at Screening
* Positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV) 1 and/or -2 antibodies at Screening.
* Excessive use of caffeine-containing beverages
* Urinary cotinine level indicative of smoking or history or regular use of tobacco- or nicotine containing products within 6 months before screening.
* History of regular alcohol consumption within 6 months of screening 10.
* Positive screen for drugs-of-abuse or cotinine.
* Blood donation in excess of 500mL within 3 months.
* Participation in another study with an experimental drug within 3 months of first IMP administration.
* Exposure to more than 4 new chemical entities within 12 months before the first IMP administration.
* Ongoing rhinitis that requires treatment.
* Use of live vaccine 28 days before dosing with study drug until telephone follow-up and use of killed vaccine 14 days before dosing with study drug until telephone follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with TEAEs and number of events will be summarised by treatment | 21 days
  Treatment Emergent Adverse Events after single and multiple dose administration will be collected at baseline and repeated until study completion

SECONDARY OUTCOMES:
Number of subjects with clinically significant abnormal haematology variables will be summarised by treatment. | 14 days
  Haemoglobin, haematocrit, MCV, MCH, MCHC, RBC, WBC and differentials will be collected at baseline and after single and multiple dose administration and repeated until Day 14.
Number of subjects with clinically significant abnormal clinical chemistry variables will be summarised by treatment. | 14 days
  Creatinine, glucose, triglycerides, urea, uric acid, bilirubin, cholesterol, sodium, potassium, alkaline phosphatase, AST, ALT and GGT will be collected at baseline and after single and multiple dose administration and repeated until Day 14.
Number of subjects with clinically significant abnormal electrocardiogram variables will be summarised by treatment. | 14 days
  RR-interval, PR (PQ)-interval, QRS-duration, QT-interval, QTcB, QTcF and heart rate will be collected at baseline and after single and multiple dose administration and repeated until Day 14.
Number of subjects with clinically significant abnormal vital sign variables will be summarised by treatment. | 14 days
  Blood pressure, pulse rate, oral body temperature and respiration rate will be collected at baseline and after single and multiple dose administration and repeated until Day 14.
Pharmacokinetics of PIN201104: The maximum observed plasma concentration (Cmax) | 24 hours
  Cmax will be calculated after single and multiple IV dosing and single SC dosing of PIN201104
PK of PIN201104: The time to reach Cmax (Tmax) | 24 hours
  Tmax will be calculated after single and multiple IV dosing and single SC dosing of PIN201104
PK of PIN201104: Apparent terminal elimination half life in plasma (t1/2) | 24 hours
  t1/2 will be calculated after single and multiple IV dosing and single SC dosing of PIN201104
PK of PIN201104: Area under the curve from time zero to the last quantifiable concentration of PIN201104 (AUC0-t) | 24 hours
  AUC0-t will be calculated after single and multiple IV dosing and single SC dosing of PIN201104
PK of PIN201104: Apparent plasma clearance of PIN201104 (CL/F) | 24 hours
  CL/F will be calculated after single and multiple IV dosing and single SC dosing of PIN201104
PK of PIN201104: Apparent volume of distribution (Vz/F) | 24 hours
  Vz/F will be calculated after single and multiple IV dosing and single SC dosing of PIN201104

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, Principal Investigator — Parexel
Locations (1):
- Investigator Site, Harrow, United Kingdom